CLINICAL TRIAL: NCT06095895
Title: Model Informed preciSion doSIng tO iNdividualise and Optimize Pharmacotherapeutic Treatment
Acronym: MISSION
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL85390.091.23
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Pharmacokinetics; Area Under Curve; Tacrolimus; Immunosuppressive Agents; Mycophenolic Acid
MeSH Terms: interventions — Phlebotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: venipuncture — An additional measurement of exposure of mycophenolic acid and/or tacrolimus will be performed

SUMMARY:
This is a prospective observational study of MIPD in clinical practice for paediatric kidney transplant patients using tacrolimus and mycophenolic acid in Radboudumc. Dose individualization in paediatric kidney transplant patients using the InsightRX platform is performed as standard care, meaning that a pharmacokinetic model and drug levels measured at t=0, t=1 and t=2 hours will be used to calculate the exposure. Based on the estimated exposure, the pharmacist gives a dose recommendation to the physician, who can then modify the dosage of mycophenolic acid or tacrolimus. The selected dose and the measured MPA and tacrolimus concentrations will be used to predict the future exposure. A second exposure measurement will be performed to evaluate whether our model is able to predict future exposure.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant patients using tacrolimus and/or mycophenolic acid
* Age between 0 and 18 years
* Indication for an AUC measurement - judgement of clinician

Exclusion Criteria:

* Incapacitated patients
* No informed consent
* Not proficient in the Dutch language

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Paediatric kidney transplant patients from Radboudumc using tacrolimus and/or mycophenolic acid.
  We will collect data for one year, in this period we expect to include 30 patients.
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2025-11-20 (Actual)

PRIMARY OUTCOMES:
Bias | 1 year
  Mean prediction error
Precision | 1 year
  Root mean squared error

CONTACTS AND LOCATIONS:
Overall Officials: Nynke Jager, Dr, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands